CLINICAL TRIAL: NCT06875934
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study Evaluating the Efficacy and Safety of SHR-1139 Injection in Patients With Moderate-to-severe Plaque Psoriasis
Brief Title: A Trial Comparing SHR-1139 Injection With Placebo in Patients With Moderate-to-severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1139-201
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1139 injection group (Experimental)
  Interventions: Drug: SHR-1139 Injection
- SHR-1139 injection placebo group (Placebo Comparator)
  Interventions: Drug: SHR-1139 Injection Placebo

INTERVENTIONS:
Drug: SHR-1139 Injection — SHR-1139 injection.
  Arms: SHR-1139 injection group
Drug: SHR-1139 Injection Placebo — SHR-1139 injection placebo.
  Arms: SHR-1139 injection placebo group

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, pharmacokinetics (PK) and immunogenicity of SHR-1139 injection in patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years old at the time of signing the informed consent form (ICF).
2. Subjects voluntarily sign informed consent form (ICF) prior to the commencement of any procedures related to the study, are able to communicate smoothly with the investigator, understand and are willing to complete the study in strict compliance with the requirements of this clinical study protocol.
3. A fertile female subject or a male subject whose partner is a fertile woman who has not had a child, has a sperm/egg donation plan for 72 weeks from the date of signing the informed consent form to the last dose, and is voluntarily using highly effective contraception (including the partner).
4. Female subjects must have negative pregnancy test results during the screening period and before randomized administration, and must be non-lactating.

Exclusion Criteria:

1. There are other skin problems that researchers believe can interfere with the evaluation of psoriasis.
2. A history of moderate to severe congestive heart failure, cardiovascular and cerebrovascular events or severe bleeding events occurred in the 3 months before screening, and the investigator considered this subject to be unfit for clinical study.
3. Had an opportunistic infection within 6 months prior to screening.
4. Allergic to the ingredients or excipients of the study drug.
5. The investigator determined that there were conditions that affected the safety and efficacy evaluation of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with at least 90% improvement (PASI 90) in their PASI (Psoriasis Area and Severity Index) score from the baseline. | At week 16.

SECONDARY OUTCOMES:
Proportion of subjects with at least 75% improvement (PASI 75) in their PASI (Psoriasis Area and Severity Index) score from the baseline. | At week 16.
Proportion of subjects with at least 100% improvement (PASI 100) in their PASI (Psoriasis Area and Severity Index) score from the baseline. | At week 16.
Adverse events (AEs) | Up to week 64.
Serum concentration of SHR-1139. | Up to week 64.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided